CLINICAL TRIAL: NCT00995514
Title: Genotype Guided Comparison of Clopidogrel and Prasugrel Outcomes Study
Acronym: GeCCO
Status: Terminated | Type: Observational
Why Stopped: Administrative reasons
Sponsor: Medco Health Solutions, Inc. (Industry)
Responsible Party: Principal Investigator, Eric Stanek, Vice President, Research, Medco Health Solutions, Inc.
Other Study IDs: GeCCO1
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Cardiovascular Disease
Keywords: acute coronary syndrome; cardiovascular death; non-fatal MI; non-fatal stroke; genetic testing; CYP2C19; clopidogrel; prasugrel; antiplatelet therapy; genotyping; bleeding
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clopidogrel: Patients receiving clopidogrel 75 mg/day as prescribed by their physician, and are extensive metabolizers by CYP2C19 genotype
- Prasugrel: Patients receiving prasugrel 5 or 10 mg/day as prescribed by their physician

SUMMARY:
The primary objective of this trial is to demonstrate the non-inferiority of clopidogrel compared to prasugrel over 6 months in cardiovascular disease patients when the clopidogrel cohort is limited to the estimated 70% of the population that are CYP2C19 extensive metabolizers. This protocol will examine the comparative effectiveness of these two strategies.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open-label, non-inferiority comparative effectiveness outcomes trial comparing clopidogrel EMs (confirmed by CYP2C19 genotype)and receiving clopidogrel at 75 mg/day with subjects receiving prasugrel at 5 and/or 10 mg/day. The antiplatelet drug clopidogrel is a commonly prescribed therapy in patients following ACS, stroke, PCI with or without stent placement, and in patients with peripheral artery disease. However, recent research suggests that in vitro anti-platelet response to clopidogrel may be limited or lost in up to 30% of treated individuals, and may be associated with inferior clinical outcomes.

The antiplatelet effect of clopidogrel requires conversion of the parent compound to an active thiol. This active thiol metabolite inhibits adenosine diphosphate (ADP)-induced platelet aggregation by blocking the platelet P2Y12 receptor, resulting in a reduction of ADP-mediated platelet aggregation. Conversion of clopidogrel to its active metabolite is a relatively inefficient process during which 85% of the pro-drug is converted to an inactive metabolite by esterases, and the remaining 15% is oxidized to the active form by cytochrome P-450 (CYP) enzymes.

The variability of clopidogrel response is associated with variability in CYP enzyme genetic expression and activity, primarily CYP2C19 which is principally responsible for the conversion of clopidogrel into its active metabolite. CYP2C19 is genetically polymorphic, with alleles that produce both reduced and enhanced drug metabolism. These polymorphisms include the loss-of-function alleles CYP2C19 *2, *3,*4 and *5 and the ultra-rapid metabolizer CYP2C19 *17.

Subjects carrying the wild-type allele for CYP2C19 (*1/*1 or extensive metabolizers, EM) are able to efficiently metabolize clopidogrel and have the greatest exposure to the active metabolite, as well as the highest levels of platelet inhibition following clopidogrel exposure. Intermediate metabolizers (IM), those individuals carrying one reduced function allele (e.g.*1/*2, *1/*3, etc), have their circulating active drug metabolite level reduced by over 30% compared to EMs resulting in a 25% reduction in platelet inhibition. These results are consistent with other studies also demonstrating that individuals carrying the CYP2C19*2 allele have decreased levels platelet aggregation inhibition following clopidogrel administration as compared to the *1/*1 wild type.

A series of recent articles have explored the effect of genetic polymorphisms in CYP2C19 on the anti-platelet activity of clopidogrel as well as clinical outcomes following PCI. Collett, et al. examined 259 patients <45 years of age who were treated with clopidogrel following a MI. Carriers for the CYP2C19*2 allele had an increased incidence of death, MI and urgent coronary revascularization (p=0.0005, HR = 3.69). Simon, et al. examined 2,208 patients that presented with acute MI and received clopidogrel therapy and found individuals that carried one or more CYP2C19 loss-of-function allele(s) had higher rates of cardiovascular events than non-carriers. The risk of death, non-fatal MI or cardiovascular stroke at 1 year after PCI was 3.58 times greater in patients carrying two loss-of-function alleles compared to wild-type patients. Trenk, et al., associated elevated platelet activity and poor clinical outcomes in patients with the*2 allele in 797 patients followed for one year after PCI.

Prasugrel is a third generation thienopyridine, and appears to have increased antiplatelet efficacy compared to clopidogrel. Like clopidogrel, prasugrel is a pro-drug that requires metabolic activation. However, esterases that are known to inactivate clopidogrel act on prasugrel to prime it for activation by a single CYP-dependant oxidation step. This more direct pathway results in a more efficient activation pathway of prasugrel.

The efficacy of prasugrel and clopidogrel have been compared head-to-head in the TRITON-TIMI 38 study. This trial enrolled 13,608 ACS patients scheduled for PCI and compared prasugrel (60-mg loading dose and then 10-mg daily maintenance dose) against clopidogrel (300-mg/75-mg), both in combination with aspirin. Results indicated that prasugrel reduced the combined rate of death from cardiovascular causes, nonfatal myocardial infarction, or nonfatal stroke (12.1% for clopidogrel vs. 9.9% for prasugrel) at 15 months post-ACS. These favorable effects on cardiovascular events were offset by an increased rate of serious bleeding (1.4%, vs. 0.9% in the clopidogrel group) and fatal bleeding (0.4% vs. 0.1%). Overall mortality did not differ between the two treatment groups.

A genetic substudy subsequently published by Mega, et al. examined the association between CYP2C19 genotypes and cardiovascular outcome in a subset of 1,477 clopidogrel-treated subjects enrolled in the TRITON-TIMI 38 study. This study demonstrated that carriers of one or more reduced-function CYP2C19 alleles had a 53% increase in the composite primary efficacy outcome compared with non-carriers (12.1% vs 8.0%, p=0.01) over 15 months of follow-up. In contrast, outcomes in a subset of prasugrel-treated patients were similar across CYP2C19 genotypes. Unfortunately, the in-trial response to clopidogrel among the genetic substudy participants differed from that of the overall clopidogrel study cohort, thus preventing direct comparisons of clopidogrel to prasugrel as a function of CYP2C19 genotype

On March 12, 2010 the FDA added a Boxed Warning to the Plavix prescribing information. The Boxed Warning concerns patients who do not effectively metabolize the drug (i.e. "poor metabolizers") and therefore may not receive the full benefits of the drug. This label modification affirms the impact of the CYP2C19 genotype on the pharmacokinetics of clopidogrel's active metabolite and, most importantly, confirmed the effect of reduced anti-platelet response with a higher rate of cardiovascular events in IM and PM populations. The event rate for clopidogrel extensive metabolizers alone has never been directly compared to prasugrel.

Upon review of data extracted from Medco's integrated claims database, the "real-world" prescribing practice of physicians for Plavix and Effient varies significantly from the narrow indication of ACS studied in the TRITON-TIMI 38 study, and from the current Effient approved labeling. Only 27% of patients new to Plavix therapy have experienced an ACS event within 6 months of the new prescription. Similarly, only 13% of new Effient users have evidence of an ACS event within 6 months of a new prescription for that agent. Overall, approximately ½ of all new Plavix users and over 80% of new Effient users have no evidence of any hospitalization event for ACS, stroke, percutaneous coronary intervention, or peripheral arterial disease, indicating that instead they have stable cardiovascular disease.

These data justify expanding the entry criteria for the GeCCO study to include patients with a recent prescription for clopidogrel or prasugrel but without a precipitating ACS event. The purpose of this study is to compare outcomes of cardiovascular disease patients prescribed Plavix or Effient in a real-world population. If, as is the case here, the population receiving these drugs includes significant numbers of patients either without recent hospitalization for ACS and/or with stable coronary disease, then the population of the GeCCO study may justifiably be expanded to include these new indications. This will afford the opportunity to fulfill its comparative effectiveness research intent through investigation of outcomes on these therapies as they are being utilized by physicians in the clinic setting.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 years and 75 years of age
* Recent prescription for clopidogrel or prasugrel.
* Participant is willing and able to provide informed consent.

Exclusion Criteria:

* Previous use of any thienopyridine within 4 months of initiating new clopidogrel or prasugrel therapy.
* Participant refusal to participate in the study.
* Anticipated discontinuation of clopidogrel or prasugrel within the 6 month study follow-up period
* Participants that have previously stated "do not contact"

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between the ages of 18 and 75 with newly initiated clopidogrel (Plavix) or prasugrel (Effient) therapy.
Sampling Method: Non-Probability Sample
Enrollment: 4471 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of clopidogrel therapy in CYP2C19 extensive metabolizers with cardiovascular disease | 6 months
  To assess the non-inferiority of clopidogrel therapy in patients with cardiovascular disease who are CYP2C19 extensive metabolizers (identified by genetic testing) compared to prasugrel therapy (non-genotyped) on the composite primary end point of cardiovascular death, hospitalization for acute coronary syndrome (nonfatal MI or unstable angina), nonfatal stroke or coronary revascularization

SECONDARY OUTCOMES:
Incidence between the two study groups of all individual components of the primary end point. | 6 and 12 months
  * Number of hospitalizations and ER visits for other cardiovascular events not included in the primary composite endpoint.
  * the primary (composite) endpoint and the individual components of the primary end point in subjects who are CYP2C19 intermediate metabolizers (IM) with clopidogrel EM and prasugrel populations
  * the primary (composite) endpoint and the individual components of the primary end point in the population of CYP2C19 intermediate and extensive metabolizers with the prasugrel population.
Total health care resource utilization and cost-effectiveness | 6 and 12 months
Health-related quality of life and activity/work productivity | 6 and 12 months
Incidence of hospitalization for site- and cause-specific bleeding | 6 and 12 months
Incidence of new or recurrent cancer | 6 and 12 months
To compare the incidence of the composite primary endpoint between the two study groups. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Stanek, Pharm.D., Principal Investigator — Medco Health Solutions, Inc.
Locations (1):
- Medco Health Solutions, Inc, Franklin Lakes, New Jersey, United States

REFERENCES:
- [Background] Collet JP, Hulot JS, Pena A, Villard E, Esteve JB, Silvain J, Payot L, Brugier D, Cayla G, Beygui F, Bensimon G, Funck-Brentano C, Montalescot G. Cytochrome P450 2C19 polymorphism in young patients treated with clopidogrel after myocardial infarction: a cohort study. Lancet. 2009 Jan 24;373(9660):309-17. doi: 10.1016/S0140-6736(08)61845-0. Epub 2008 Dec 26. PMID 19108880
- [Background] Trenk D, Hochholzer W, Fromm MF, Chialda LE, Pahl A, Valina CM, Stratz C, Schmiebusch P, Bestehorn HP, Buttner HJ, Neumann FJ. Cytochrome P450 2C19 681G>A polymorphism and high on-clopidogrel platelet reactivity associated with adverse 1-year clinical outcome of elective percutaneous coronary intervention with drug-eluting or bare-metal stents. J Am Coll Cardiol. 2008 May 20;51(20):1925-34. doi: 10.1016/j.jacc.2007.12.056. PMID 18482659
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias W, Braunwald E, Sabatine MS. Cytochrome p-450 polymorphisms and response to clopidogrel. N Engl J Med. 2009 Jan 22;360(4):354-62. doi: 10.1056/NEJMoa0809171. Epub 2008 Dec 22. PMID 19106084
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083